CLINICAL TRIAL: NCT06642792
Title: A Phase I/II Study of AK129 (Bispecific Antibody Targeting LAG-3 and PD-1) Monotherapy or in Combination With AK117 (Anti-CD47 Monoclonal Antibody) in Relapse or Refractory Classic Hodgkin Lymphoma With PD-1/L1 Inhibitor Treatment Failure
Brief Title: A Study of AK129 With or Without AK117 in PD(L)1-refractory Classic Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK129-102
Record Dates: First submitted 2024-09-26; First posted 2024-10-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Classic Hodgkin Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK129 (Experimental): Phase Ia: Subjects will receive AK129: different doses on every 2 weeks.
  Interventions: Drug: AK129
- AK129+AK117 (Experimental): Phase Ib: Subjects will receive: AK129: different doses on every 2 weeks, AK117: 30mg/kg on every 2 weeks.
  Phase II: Subjects will receive: AK129: recommended phase II dose (RP2D) from phase Ib on every 2 weeks, AK117: 30mg/kg on every 2 weeks.
  Interventions: Drug: AK129; Drug: AK117

INTERVENTIONS:
Drug: AK129 — Subjects receive AK129 intravenously.
Drug: AK117 — Subjects receive AK117 intravenously.
  Arms: AK129+AK117

SUMMARY:
This is a phase I/II study. All subjects are patients diagnosed with relapse or refractory (R/R) classic Hodgkin lymphoma (cHL) and has progressed on treatment with PD-1/L1 inhibitor therapy. The purpose of this study is to evaluate the safety and efficacy of AK129 (bispecific antibody targeting LAG-3 and PD-1) monotherapy or in combination with AK117 (anti-CD47 monoclonal antibody) in R/R cHL with PD-1/L1 inhibitor treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at the time of enrolment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected Survival of ≥ 12 weeks.
* Diagnosed as R/R cHL according to Lugano 2014 criteria.
* Has progressed on treatment with PD-1/L1 inhibitior therapy.
* Has adequate organ function.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception from the start of screening until 120 days after the last dose of study treatment.

Exclusion Criteria:

* Diagnosed with nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL) or gray zone lymphoma.
* Central nervous system (CNS) lymphoma involvement.
* Known history of human T-cell leukemia virus type 1 (HTLV-1) infection.
* Autologous hematopoietic stem cell transplantation (auto-HSCT) or chimeric antigen receptor T cell immunotherapy (CAR-T) within 90 days prior to the first dose of study treatment.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation (allo-HSCT).
* Previous use of any agents targeting the CD47-SIRPα pathway, LAG-3 pathway, or similar targets.
* Has other malignancies within 3 years prior to the first dose or residual lesions from other malignancies diagnosed more than 3 years ago.
* Has an active autoimmune disease requiring systemic treatment within 2 years prior to the first dose.
* History of active or previously confirmed inflammatory bowel disease.
* History of interstitial lung disease requiring corticosteroid therapy, or current interstitial lung disease.
* Has known active Hepatitis B or Hepatitis C.
* Unresolved toxicity from previous anti-tumor treatment.
* Uncontrolled comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Phase I: Number of participants with dose limiting toxicity (DLT) | Within the first 28 days following the first dose of study treatment.
  Any untoward medical occurrence in a subject within the first 28 days following the first dose, considered related to the study treatment.
Phase I/II: Incidence and severity of adverse events (AEs) | Up to approximately 2 years.
  Any untoward medical occurrence in a subject, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Phase I/II: Objective response rate (ORR) | Up to approximately 2 years
  The proportion of subjects achieving complete response (CR) or partial response (PR) assessed by investigator per Lugano 2014 criteria.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  The proportion of subjects achieving complete response (CR) , partial response (PR) or stable disease (SD) assessed by investigator per Lugano 2014 criteria.
Time to response (TTR) | Up to approximately 2 years
  The time from cycle 1 day 1(C1D1) to the first recorded response assessed by investigator per Lugano 2014 criteria.
Duration of response (DoR) | Up to approximately 2 years
  The time from the first recorded response until disease progression assessed by investigator or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to approximately 2 years
  The time from C1D1 until disease progression assessed by investigator or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to approximately 2 years
  The time from C1D1 until death due to any cause.
Maximum concentration (Cmax) | Up to approximately 2 years
  The maximum concentration of the drug observed in the blood plasma after administration.
Time to maximum concentration (Tmax) | Up to approximately 2 years
  The time taken to reach the maximum concentration (Cmax) of the drug in the blood plasma.
Area under the curve (AUC) | Up to approximately 2 years
  The area under the plasma concentration versus time curve, which represents the total drug exposure over time.
Half-life (T1/2) | Up to approximately 2 years
  The time required for the plasma concentration of the drug to decrease by half.
Anti-drug antibody (ADA) | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Wenting Li, MD, Study Director — Akeso
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No